CLINICAL TRIAL: NCT02097901
Title: Microfracture in Rotator Cuff Injury Repair
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient patient material
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Morten S. Wad, M.D, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJ-370
Record Dates: First submitted 2014-03-17; First posted 2014-03-27 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Rupture of the Rotator Cuff
Keywords: Rotator Cuff; Injury; Repair; Microfracture; Healing
MeSH Terms: conditions — Wounds and Injuries; Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Microfracture (Experimental): Rotator Cuff Repair AND Microfracture at rotatorcuff footprint
  Interventions: Procedure: Microfracture
- NO microfracture (Active Comparator): Rotator cuff reinsertion without microfracture
  Interventions: Procedure: NO microfracture

INTERVENTIONS:
Procedure: Microfracture — Rotator Cuff Repair AND Microfracture
  Arms: Microfracture
Procedure: NO microfracture — Rotator Cuff Repair without microfracture
  Arms: NO microfracture

SUMMARY:
The hypothesis is that microfractures in the footprint of the humerus will aid to improve the tendon healing to the bone. The aim of the study is to investigate whether the use of microfractures at the footprint of the rotator cuff will improve the tendon healing when reinserted. Patients undergoing surgery for a rotator cuff injury will be randomised to repair with or without microfracture.

ELIGIBILITY:
Inclusion Criteria:

- Patients over the age of 18 with a full thickness rotatorcuff rupture.

Exclusion Criteria:

* Isolated rupture of the subscapularis
* Tendon atrophia
* Goutallier grade 3-4 fatty degeneration
* Fracture surgery in same shoulder
* Inflammatory or neurologic affection of shoulder
* Other disabling disease
* Unwilling to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change in Western Ontario Rotator Cuff Index (WORC) | 0, 3 and 12 months
  Standardized questionnaire
Change in Quick Disabilities of the Arm, Shoulder and Hand (Quick-DASH) | 0, 3 and 12 months
  Standardized questionnaire

SECONDARY OUTCOMES:
MRI integrity of the rotatorcuff | 12 months
  * Intact rotatorcuff
  * Partial rupture
  * Full thickness rupture

OTHER OUTCOMES:
Strength of rotatorcuff | 3 and 12 months
  Strength 0-5 in abduction and external rotation.
Function of rotatorcuff | 3 and 12 months
  Range of movement in abduction and external rotation in full degrees.
Complications | 12 months
  Assesses the complication rate in each group such as infection, bleeding and reoperation.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Blønd, M.D, Study Director — Køge Sygehus; Gunner S Barfoed, M.D, Study Director — Køge Sygehus; Thomas JN Sørensen, M.D, Study Director — Køge Sygehus
Locations (1):
- Køge Sygehus, Køge, Lykkebækvej 1, Denmark